CLINICAL TRIAL: NCT05032859
Title: A Phase 3 Efficacy and Safety Study of Tapinarof for the Treatment of Moderate to Severe Atopic Dermatitis in Children and Adults
Brief Title: Tapinarof for the Treatment of Atopic Dermatitis in Children and Adults (DMVT-505-3102)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMVT-505-3102
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
Keywords: eczema; pediatric; tapinarof; phase 3; topical
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Intervention Model Description: Following a 30-day screening period, eligible subjects will be randomized at a 2:1 ratio to receive once daily treatment with tapinarof cream, 1% or vehicle cream.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, study center staff, subject, and sponsor will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- tapinarof cream (Experimental): tapinarof cream, 1%, applied topically once daily
  Interventions: Drug: tapinarof cream, 1%
- vehicle cream (Placebo Comparator): vehicle cream, applied topically once daily
  Interventions: Drug: vehicle cream

INTERVENTIONS:
Drug: tapinarof cream, 1% — applied topically once daily
  Arms: tapinarof cream
Drug: vehicle cream — applied topically once daily
  Arms: vehicle cream

SUMMARY:
This is a double-blind, randomized, vehicle controlled Phase 3 study to evaluate the efficacy and safety of topical tapinarof cream, 1% compared to vehicle control cream in pediatric and adult subjects with atopic dermatitis.

DETAILED DESCRIPTION:
This study is a 8-week double-blind, vehicle-controlled treatment study in which subjects will be randomized to receive tapinarof cream, 1% or vehicle cream once daily for 8 weeks. At the end of the 8-week study treatment, qualified subjects will have the option to enroll in an open-label, long-term extension study for an additional 48 weeks of treatment. Subjects who do not participate in the open-label, long-term extension study will complete a follow-up visit approximately one week after the end of treatment in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 2 and above with clinical diagnosis of AD
* Subject with atopic dermatitis covering ≥5% and ≤ 35% of the BSA
* A vIGA-AD score of ≥3 at screening and baseline
* An EASI score of ≥6 at screening and baseline
* Atopic dermatitis present for at least 6 months for ages 6 years old and above or 3 months for ages 2 to 5 years old
* Female subjects of childbearing potential who are engaging in sexual activity that could lead to pregnancy should use acceptable birth control methods
* Must not be pregnant
* Subject, subject's parent, or legal representative must be capable of giving written informed consent/assent

Exclusion Criteria:

* Immunocompromised at screening
* Chronic or acute systemic or superficial infection requiring treatment with systemic antibacterials or antifungals within one week prior to baseline visit
* Significant dermatological or inflammatory condition other than AD that, in the Investigator's opinion, would make it difficult to interpret data or assessments during the study
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2.0x the upper limit of normal (ULN).
* Screening total bilirubin > 1.5x ULN
* Current or chronic history of liver disease
* Current or history of cancer within 5 years except for adequately treated cutaneous basal cell carcinoma, squamous cell carcinoma or carcinoma in situ of the cervix
* Subjects who would not be considered suitable for topical therapy
* Use of any prohibited medication or procedure within the indicated period before the baseline visit including other investigational product within 30 days or 5 half-lives of the investigational product (whichever is longer)
* History of or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the Investigator's opinion, may interfere with the subject's participation in the study, interpretation of results, or ability to understand and give informed consent.
* Pregnant or lactating females
* History of sensitivity to the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the -Investigator or Medical Monitor, contraindicates their participation
* Previous known participation in a clinical study with tapinarof (previously known as GSK2894512 and WBI-1001)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Villalobos, Study Director — Dermavant Sciences, Inc.
Locations (57):
- United States (52):
  - Dermavant Investigative Site, Birmingham, Alabama
  - Dermavant Investigative Site, Scottsdale, Arizona
  - Dermavant Investigative Site, Fort Smith, Arkansas
  - Dermavant Investigative Site, Cerritos, California
  - Dermavant Investigative Site, Huntington Beach, California
  - Dermavant Investigative Site, Lancaster, California
  - Dermavant Investigative Site, Long Beach, California
  - Dermavant Investigative Site, Los Angeles, California
  - Dermavant Investigative Site, San Diego, California
  - Dermavant Investigative Site, San Francisco, California
  - Dermavant Investigative Site, Santa Ana, California
  - Dermavant Investigative Site, Santa Monica, California
  - Dermavant Investigative Site, Boca Raton, Florida
  - Dermavant Investigative Site, Delray Beach, Florida
  - Dermavant Investigative Site, Jacksonville, Florida
  - Dermavant Investigative Site, Miami, Florida
  - Dermavant Investigative Site, Miami Lakes, Florida
  - Dermavant Investigative Site, Tampa, Florida
  - Dermavant Investigative Site, Snellville, Georgia
  - Dermavant Investigative Site, Evansville, Indiana
  - Dermavant Investigative Site, Overland Park, Kansas
  - Dermavant Investigative Site, Lexington, Kentucky
  - Dermavant Investigative Site, Louisville, Kentucky
  - Dermavant Investigative Site, Baton Rouge, Louisiana
  - Dermavant Investigative Site, New Orleans, Louisiana
  - Dermavant Investigative Site, Rockville, Maryland
  - Dermavant Investigative Site, Detroit, Michigan
  - Dermavant Investigative Site, Lincoln, Nebraska
  - Dermavant Investigative Site, Omaha, Nebraska
  - Dermavant Investigative Site, Las Vegas, Nevada
  - Dermavant Investigative Site, East Windsor, New Jersey
  - Dermanvant Investigative Site, Brooklyn, New York
  - Dermavant Investigative Site, Watertown, New York
  - Dermavant Investigative Site, Charlotte, North Carolina
  - Dermavant Investigative Site, Dayton, Ohio
  - Dermavant Investigative Site, Mason, Ohio
  - Dermavant Investigative Site, Mayfield Heights, Ohio
  - Dermavant Investigative Site, Tulsa, Oklahoma
  - Dermavant Investigative Site, Medford, Oregon
  - Dermavant Investigative Site, Portland, Oregon
  - Dermavant Investigative Site, East Greenwich, Rhode Island
  - Dermavant Investigative Site, Anderson, South Carolina
  - Dermavant Investigative Site, North Charleston, South Carolina
  - Dermavant Investigative Site, Spartanburg, South Carolina
  - Dermavant Investigative Site, Memphis, Tennessee
  - Dermavant Investigative Site, Bellaire, Texas
  - Dermavant Investigative Site, Dripping Springs, Texas
  - Dermavant Investigative Site, Grapevine, Texas
  - Dermavant Investigative Site, Houston, Texas
  - Dermavant Investigative Site, San Antonio, Texas
  - Dermavant Investigative Site, Webster, Texas
  - Dermavant Investigative Site, Spokane, Washington
- Canada (5):
  - Dermavant Investigative Site, Surrey, British Columbia
  - Dermavant Investigative Site, Barrie, Ontario
  - Dermavant Investigative Site, Markham, Ontario
  - Dermavant Investigative Site, Waterloo, Ontario
  - Dermavant Investigative Site, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silverberg JI, Eichenfield LF, Hebert AA, Simpson EL, Stein Gold L, Bissonnette R, Papp KA, Browning J, Kwong P, Korman NJ, Brown PM, Rubenstein DS, Piscitelli SC, Somerville MC, Tallman AM, Kircik L. Tapinarof cream 1% once daily: Significant efficacy in the treatment of moderate to severe atopic dermatitis in adults and children down to 2 years of age in the pivotal phase 3 ADORING trials. J Am Acad Dermatol. 2024 Sep;91(3):457-465. doi: 10.1016/j.jaad.2024.05.023. Epub 2024 May 20. PMID 38777187
- [Derived] Alexis AF, Kircik L, Chovatiya R, Rice ZP, Soong W, Bhutani T, Brown PM, Piscitelli SC, Rubenstein DS, Tallman AM, Armstrong AW. Tapinarof Cream for Adults and Children with Atopic Dermatitis-Efficacy by Race and Fitzpatrick Skin Type in Two Phase 3 Randomized Clinical Trials. Dermatol Ther (Heidelb). 2025 Sep;15(9):2667-2682. doi: 10.1007/s13555-025-01489-w. Epub 2025 Jul 22. PMID 40696240
- [Derived] Gold LS, Bruno MJ, Lewitt GM, Hebert AA. Characteristics and management of follicular events and contact dermatitis in patients using tapinarof cream for the treatment of atopic dermatitis or plaque psoriasis. J Dermatolog Treat. 2025 Dec;36(1):2517388. doi: 10.1080/09546634.2025.2517388. Epub 2025 Jul 2. PMID 40600584
- [Derived] Gold LS, Del Rosso J, Ehst BD, Zirwas MJ, Green LJ, Brown PM, Rubenstein DS, Piscitelli SC, Tallman AM. Tapinarof cream 1% once daily was well tolerated in adults and children with atopic dermatitis in two phase 3 randomized trials. J Dermatolog Treat. 2025 Dec;36(1):2444489. doi: 10.1080/09546634.2024.2444489. Epub 2025 Jan 12. PMID 39799945
- [Derived] Simpson EL, Hebert AA, Browning J, Serrao RT, Sofen H, Brown PM, Piscitelli SC, Rubenstein DS, Tallman AM. Tapinarof Improved Outcomes and Sleep for Patients and Families in Two Phase 3 Atopic Dermatitis Trials in Adults and Children. Dermatol Ther (Heidelb). 2025 Jan;15(1):111-124. doi: 10.1007/s13555-024-01318-6. Epub 2025 Jan 7. PMID 39777610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from the main study (DMVT-505-3102) had the option to participate in the open label extension study (DMVT-505-3103, NCT05142774).
Period: Overall Study
Arm/Group | Tapinarof Cream | Vehicle Cream
Started | 271 | 135
Completed | 235 | 106
Not Completed | 36 | 29

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapinarof Cream | Vehicle Cream | Total
Number analyzed (Participants) | 271 | 135 | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.4 (16.24) | 16.7 (16.05) | 16.5 (16.16)
Age, Customized [Count of Participants; unit: Participants]
  2-6 Years | 65 | 32 | 97
  7-11 Years | 64 | 32 | 96
  12-17 Years | 89 | 44 | 133
  ≥18 Years | 53 | 27 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 77 | 231
  Male | 117 | 58 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 27 | 76
  Not Hispanic or Latino | 221 | 107 | 328
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 39 | 23 | 62
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 95 | 47 | 142
  White | 124 | 58 | 182
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Number; unit: Count of participants]
  Canada | 41 | 22 | 63
  United States | 230 | 113 | 343
Validated Investigator Global Assessment for Atopic Dermatitis [Count of Participants; unit: Participants] — Grading (per protocol score definition):
  * 0: Clear - No inflammatory signs of atopic dermatitis.
  * 1: Almost Clear - Barely perceptible erythema, induration/papulation, and/or minimal lichenification.
  * 2: Mild - Slight but definite erythema (pink), slight but definite induration/papulation, and/or slight but definite lichenification.
  * 3: Moderate - Clearly perceptible erythema (dull red), clearly perceptible induration/papulation, and/or clearly perceptible lichenification.
  * 4: Severe - Marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification.
  Participants
    0 - Clear | 0 | 0 | 0
    1 - Almost Clear | 0 | 0 | 0
    2 - Mild | 0 | 0 | 0
    3 - Moderate | 228 | 113 | 341
    4 - Severe | 43 | 22 | 65
Percent Body Surface Area (BSA) [Mean (Standard Deviation); unit: Percentage of Affected BSA] | 17.13 (8.743) | 15.84 (7.888) | 16.70 (8.480)
Eczema Area and Severity Index (EASI) [Mean (Standard Deviation); unit: units on a scale] | 13.45 (5.615) | 13.09 (4.689) | 13.33 (5.322)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Who Have a Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) Score of Clear or Almost Clear (0 or 1) With a Minimum 2-grade Improvement From Baseline to Week 8. Analyses Were Done Using Multiple Imputation.
Description: The vIGA-AD is a global assessment of the current state of the disease. It is a static 5-point scale used to grade overall disease severity (scalp excluded), as determined by the investigator, using the clinical characteristics of erythema, induration/papulation, lichenification, oozing/crusting. The vIGA-AD ranges from 0 to 4 and is calculated as Clear (0), Almost clear (1), Mild (2), Moderate (3), and Severe (4). Higher vIGA-AD scores represent more severe disease.
  Statistics are based on 100 imputed datasets.
Time Frame: Baseline to Week 8
Population: ITT Population (MI Estimand)
Measure: Number; unit: Percentage of participants
Arm/Group | Tapinarof Cream | Vehicle Cream
Number analyzed (Participants) | 271 | 135
Percentage of participants | 46.4 | 18.0
Statistical Analysis 1: Comparison: Tapinarof Cream vs Vehicle Cream; H0: The proportion of subjects who achieve a vIGA-AD score of clear (0) or almost clear (1) and at least a 2-grade reduction from Baseline at Week 8 is equal between tapinarof cream, 1% and vehicle cream; H1: The proportion of subjects who achieve a vIGA-AD score of clear (0) or almost clear (1) and at least a 2-grade reduction from Baseline at Week 8 is different between the tapinarof cream, 1% and vehicle cream; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by Baseline vIGA-AD Score and Age Group; Risk Ratio, log = 2.27, 95% CI 2-sided [1.54 to 3.32] — Adjusted logit-based estimate of the common relative risk of success (Tapinarof Cream 1%/Vehicle Cream) over all strata. Multiple imputation p-value is for null hypothesis that the log (Relative Risk) equals 0

2. Secondary Outcome: Percent of Subjects With ≥ 75% Improvement in Eczema Area and Severity Index (EASI) From Baseline to Week 8. Analyses Were Done Using Multiple Imputation.
Description: The Eczema Area and Severity Index (EASI) is a scoring system that takes into account the overall severity of disease based on lesion severity and the extent of percent body surface area affected with atopic dermatitis. The EASI is a composite score ranging from 0 -72 that takes into account the degree of erythema, edema/papulation, excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the percent body surface area involved for each body region relative to the whole body. A higher EASI score represents more severe disease.
  Statistics are based on 100 imputed datasets.
Time Frame: Baseline to Week 8
Population: ITT Population (MI Estimand)
Measure: Number; unit: Percentage of participants
Arm/Group | Tapinarof Cream | Vehicle Cream
Number analyzed (Participants) | 271 | 135
Percentage of participants | 59.1 | 21.2
Statistical Analysis 1: Comparison: Tapinarof Cream vs Vehicle Cream; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by vIGA-AD score at Baseline (vIGA-AD scores of 3 or 4) and age group (2-6 yrs, 7-11 yrs, 12-17 yrs, 18+ yrs); Risk Ratio, log = 2.14, 95% CI 2-sided [1.53 to 3.00] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Change in in Percent of Total Body Surface Area (%BSA) Affected From Baseline to Week 8.
Description: Assessment of percent body surface area (%BSA) is an estimate of the percentage of total involved skin with atopic dermatitis. Estimates were made using the handprint method, where the full palmar hand of the participant (fully extended palm, fingers and thumbs together) represented approximately 1% of the total BSA. Body regions are assigned a specific number of handprints with associated percentages (Head and neck = 10% [10 handprints], upper extremities = 20% [20 handprints], trunk (including axillae and groin) = 30% [30 handprints], lower extremities, including buttocks, = 40% [40 handprints]). Estimates of the percent involvement of each body region will be multiplied by the fraction of total body area to obtain the total %BSA involved by region and overall.
Time Frame: Baseline to Week 8
Population: ITT Population (MI Estimand)
Measure: Mean (Standard Error); unit: Change in affected BSA percentage
Arm/Group | Tapinarof Cream | Vehicle Cream
Number analyzed (Participants) | 271 | 135
Change in affected BSA percentage | -10.36 (0.540) | -3.14 (0.676)
Statistical Analysis 1: Comparison: Tapinarof Cream vs Vehicle Cream; Test type: Superiority; p < 0.0001, ANCOVA; age*vIGA cohort and treatment as categorical covariates, and baseline %BSA as a continuous covariate; Least squares mean difference = -6.60, 95% CI 2-sided [-8.17 to -5.02], Standard Error of Mean 0.803

4. Secondary Outcome: Percent of Subjects With ≥ 90% Improvement in Eczema Area and Severity Index (EASI) From Baseline to Week 8. Analyses Were Done Using Multiple Imputation.
Description: as for outcome 2
Time Frame: Baseline to Week 8
Population: ITT Population (MI Estimand)
Measure: Number; unit: Percentage of participants
Arm/Group | Tapinarof Cream | Vehicle Cream
Number analyzed (Participants) | 271 | 135
Percentage of participants | 30.1 | 10.0
Statistical Analysis 1: Comparison: Tapinarof Cream vs Vehicle Cream; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel; Stratified by Baseline vIGA-AD Score and Age Group; Risk Ratio, log = 2.34, 95% CI 2-sided [1.39 to 3.94] — [estimate comment as in outcome 1, analysis 1]; Adjusted logit-based estimate of the common relative risk of success (Tapinarof Cream 1%/Vehicle Cream) over all strata. Multiple imputation p-value is for null hypothesis that the log (Relative Risk) equals 0

5. Secondary Outcome: Percent of Subjects ≥ 12 Years Old With a Baseline Peak Pruritis-Numeric Rating Scale (PP-NRS) Score ≥ 4 Who Achieve ≥ 4-point Reduction in the Average Weekly PP-NRS From Baseline to Week 8.
Description: The Peak Pruritus Numeric Rating Scale (PP-NRS) is used to quickly assess itch/pruritus severity over a 24-hour period. The PP-NRS is scored on a scale of 0 to 10, with 0 being "no itch" and 10 being "worst itch imaginable". The subject will utilize the scale to assess peak pruritis once per day and record the results in their diaries. The daily ratings are averaged to generate a score for the week.
  Statistics are based on 100 imputed datasets.
Time Frame: Baseline to Week 8
Population: ITT Population (MI Estimand)
Measure: Number; unit: Percentage of participants
Arm/Group | Tapinarof Cream | Vehicle Cream
Number analyzed (Participants) | 271 | 135
Percentage of participants | 52.8 | 24.1
Statistical Analysis 1: Comparison: Tapinarof Cream vs Vehicle Cream; Test type: Superiority; p = 0.0015, Cochran-Mantel-Haenszel; Stratified by Baseline vIGA-AD Score and Age Group; Risk Ratio, log = 2.17, 95% CI 2-sided [1.34 to 3.50] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Through study completion, up to 9 weeks
Arm/Group | Tapinarof Cream | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/271 | 0/133
Serious Adverse Events (participants affected / at risk) | 2/271 | 0/133
Other Adverse Events (participants affected / at risk) | 55/271 | 13/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tapinarof Cream (N=271) | Vehicle Cream (N=133)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Psychogenic seizure (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tapinarof Cream (N=271) | Vehicle Cream (N=133)
Pyrexia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Folliculitis (Infections and infestations) | 22 (23) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 2 (2)
COVID-19 (Infections and infestations) | 6 (6) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (3)
Ear infection (Infections and infestations) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT05032859/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT05032859/SAP_001.pdf